CLINICAL TRIAL: NCT03942055
Title: Prospective Observational Study: The Association of B-7 Lung Ultrasound Pattern With the Development of Postoperative Pulmonary Edema After Major Non-cardiac Surgery
Brief Title: The Association of B-7 Lung Ultrasound Pattern With the Development of Postoperative Pulmonary Edema
Status: Withdrawn | Type: Observational
Why Stopped: PI determined not enough clinical staff support for project.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew Barker, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F34567890
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- B-line score ≥7: Patients with B-line score ≥7 at the end of the surgical procedure.
  The Sonosite Edge II Ultrasound device will be used.
  The B-line score will be partially based on the simplified 4-sector lung ultrasound scoring protocol used by Phillip Enghard at el. The Enghard study showed a closed correlation between the number of B-lines per intercostal space and EVLW Index measurements.
  Interventions: Device: Sonosite Edge II Ultrasound
- B-line score <7: Patients with B-line score <7 at the end of the surgical procedure.
  The Sonosite Edge II Ultrasound device will be used.
  The B-line score will be partially based on the simplified 4-sector lung ultrasound scoring protocol used by Phillip Enghard at el. The Enghard study showed a closed correlation between the number of B-lines per intercostal space and EVLW Index measurements.
  Interventions: Device: Sonosite Edge II Ultrasound

INTERVENTIONS:
Device: Sonosite Edge II Ultrasound — Certified by UAB Biomedical and Clinical Engineering Dept- certification #9365 Mechanism of Action: Point of Care Bedside Ultrasound

SUMMARY:
The objective of this proposal is to conduct a randomized controlled study to examine the association between the increase in extravascular lung water as determined by lung ultrasound and the development of radiologic pulmonary edema as diagnosed by chest roentgenogram in patients undergoing major elective open intra-peritoneal surgeries under general endotracheal anesthesia.

DETAILED DESCRIPTION:
This study will be conducted at the University of Alabama at Birmingham's post- anesthesia care unit (PACU). A total of 60 patients will be randomly selected from the 5th and 7th floor surgical suite daily display boards and enrolled in the study. A preoperative and postoperative Point of Care (POCUS) lung U/S exam and Point of Care (POCUS) transthoracic echo will be performed with a Sonosite Edge II bedside U/S machine (approved by UAB Biomedical and Clinical Engineering Dept-#9365) in the pre-anesthesia holding area before the surgical procedure, and after the end of the procedure in the post- anesthesia care unit (PACU). EVLW will be defined as B-line score ≥7 before and after the surgical procedure. Pulmonary edema will be defined by the official radiology report on a chest X ray in the first 72 hrs postoperatively. Pre and Post Op POCUS Pulmonary Capillary Wedge Pressure (PCWP) will be obtained via Trans-thoracic bedside Ultrasound measuring Mitral Valve Inflow (E) Velocity and Early Diastolic Lateral Mitral Annulus Velocity/Tissue Doppler Imaging (E'). A 5-1Mhz Phased Array Probe will be used to obtain images. The PCWP data obtained will be used to correlate with EVLW findings. Ultrasound windows for PCWP measurements will be obtained using the Apical 4-chamber View and/or modified Subcostal View.-

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age, undergoing major elective intraperitoneal surgeries expected to be in hospital for 72 hours

Exclusion Criteria:

* Patients < 18 years
* Pregnant females
* Cardiac EF 40% on last pre-operative echo
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled in a sequential manner from the Kirklin Clinic Pre-operative Anesthesia clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pulmonary Edema | 72 hours after the surgical procedure
  The development of newly onset pulmonary edema as diagnosed by chest X ray in the first 72 hrs post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Zaky, MD MPH FCCM, Study Chair — UAB Department of Anesthesiology, Critical Care Division

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jaffee W, Hodgins S, McGee WT. Tissue Edema, Fluid Balance, and Patient Outcomes in Severe Sepsis: An Organ Systems Review. J Intensive Care Med. 2018 Sep;33(9):502-509. doi: 10.1177/0885066617742832. Epub 2017 Nov 26. PMID 29172943
- [Result] Assaad S, Kratzert WB, Shelley B, Friedman MB, Perrino A Jr. Assessment of Pulmonary Edema: Principles and Practice. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):901-914. doi: 10.1053/j.jvca.2017.08.028. Epub 2017 Aug 19. PMID 29174750